CLINICAL TRIAL: NCT02045940
Title: A Randomized Double Blinded (Sponsor Unblind), Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Selective Androgen Receptor Modulator (SARM) in Single and Repeat Doses in Healthy Male Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of GSK2881078 in Single and Repeat Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200181
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Cachexia
Keywords: FTIH; pharmacokinetics; SARM; safety
MeSH Terms: conditions — Cachexia | interventions — GSK2881078

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Participants will receive one of the following four treatment sequences in four study period (one treatment per period). Sequence 1=Placebo, dose level (DL) 2, DL3, and DL4. Sequence 2=DL1, placebo, DL2, and DL4. Sequence 3=DL1, DL2, placebo, and DL4. Sequence 4=DL1, DL2, DL3, and placebo
  Interventions: Drug: GSK2881078; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive one of the following four treatment sequences in four study period (one treatment per period). Sequence 5=Placebo, DL5, DL6, and DL7. Sequence 6=DL4, placebo, DL6, and DL7. Sequence 7=DL4, DL5, placebo, and DL7. Sequence 8=DL4, DL5, DL6, and placebo
  Interventions: Drug: GSK2881078; Drug: Placebo
- Cohort 3 (Experimental): Participants will receive repeat doses of GSK2881078 or placebo in a 3:1 randomization ratio for 14 days. The dose level will depend upon results from Part A
  Interventions: Drug: GSK2881078; Drug: Placebo
- Cohort 4 (Experimental): Participants will receive repeat doses of GSK2881078 or placebo in a 3:1 randomization ratio for 14 days. The dose level will depend upon results from Part A and preceding repeat dose Cohort
  Interventions: Drug: GSK2881078; Drug: Placebo
- Cohort 5 (Experimental): Participants will receive repeat doses of GSK2881078 or placebo in a 3:1 randomization ratio for 14 days. The dose level will depend upon results from Part A and preceding repeat dose Cohorts
  Interventions: Drug: GSK2881078; Drug: Placebo

INTERVENTIONS:
Drug: GSK2881078 — Hot melt solution within Capsule for oral single ascending doses or repeat dose administration with planned dose level and strength of 0.1, 0.3, 1.0, 2.0, 4.0, 8.0, and 10.0 mg
Drug: Placebo — Hot melt solution within Capsule for oral single ascending doses or repeat doses administration.

SUMMARY:
This study is the first administration of GSK2881078 to humans. The intention of this study is to provide sufficient confidence in the safety of the molecule to inform progression to further repeat dose and proof of concept studies. This study will include approximately 52 subjects and consist of 2 parts. Part A will consist of two cohorts of 8 subjects to assess the safety, tolerability, and pharmacokinetic (PK) of ascending single oral doses of GSK2881078. Cohorts 1 and 2 will include healthy male subjects. Part B (Cohorts 3, 4 and 5) will include three cohorts of 12 healthy male subjects to examine the safety, tolerability, PK, and pharmacodynamic (PD) of repeated doses of GSK2881078 over 14 days. The total duration of the study including screening and follow-up, is not expected to exceed 70 days.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 50 years of age (inclusive), at the time of signing the informed consent form
* Body weight >= 50 kilogram (kg) and Body Mass Index (BMI) within the range 19 - 32 kg/meter square (m^2) (inclusive), where BMI= weight in kg/ height in m^2
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the Lifestyle Section of the protocol. This criterion must be followed through the completion of the follow-up visit.
* Average QTcF <450millisecond (msec); or QTcF <480msec in subjects with Bundle Branch Block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subjects with a history of clinically significant endocrine, gastrointestinal, hepatic, cardiovascular, neurological, haematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
* Subjects with a history at any time in the past of coronary artery disease, congestive heart failure, angina, myocardial infarction, any cardiac surgery, valvular heart disease, clinically significant arrhythmia, dyspnea, pulmonary edema, stroke, or transient ischemic attack. ECG exclusion criteria: Heart rate-<40 and >100 beats per minute, PR Interval-<120 and >200msec, QRS duration-<70 and >110msec.
* Subjects with a history of malignancy that is not in complete remission for at least 5 years or 1 year for non-melanoma skin carcinoma
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of drug or alcohol abuse within 5 years prior to the Screening Period.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects with a family history of early onset prostate cancer or multiple members with prostate cancer.
* A positive pre-study drug or alcohol screen.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Subjects with values outside the specified ranges for the following Key Clinical Laboratory Tests must be excluded from the study:

Liver function tests - Alanine aminotransferase, Direct Bilirubin, or Albumin more than 10% outside the normal reference range (<0.9 x lower limit of normal [LLN] or >1.1 x upper limit of normal [ULN]) Renal function - Creatinine >1.6milligrams (mg)/deciliter (dL) with an age appropriate glomerular filtration rate<=60 (mL/minute/1.73 m^2).

Electrolytes - Sodium more than ± 5milliequivalents/Liter outside the normal reference range, Potassium or Calcium more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN) Metabolic - Glucose more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN) and Total Cholesterol > 240mg/dL Muscle - creatine phosphokinase >2.0 x ULN Hematology - Hemoglobin, white blood cells, Neutrophils, or Platelets more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN) Prostate Specific Antigen >2.5nanogram/mL

* A positive test for human immuno virus antibody
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and throughout the study, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months (12 weeks), 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56-day period.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2015-03-26 (Actual); Study Completion 2015-03-26 (Actual)

PRIMARY OUTCOMES:
Vital sign assessment following single doses as a measure of safety and tolerability | Up to 61 days
  Vital signs include: systolic blood pressure, diastolic blood pressure and heart rate
Vital sign assessment following repeat doses as a measure of safety and tolerability | Up to 56 days
  Vital signs include: systolic blood pressure, diastolic blood pressure and heart rate
Cardiac telemetry following single doses as a measure of safety and tolerability | Up to 19 days
  Continuous cardiac telemetry will be performed for at least 12 hours post dose in each treatment period in Part A.
Cardiac telemetry following repeat doses as a measure of safety and tolerability | 14 days
  Continuous cardiac telemetry will be performed for at least 8 hours post dose in Days 1, 4, 7, 10, and 14 in Part B
Electrocardiogram (ECG) assessment following single doses as a measure of safety and tolerability | Up to 61 days
  12-lead ECGs will be obtained during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF intervals) at each timepoint
ECG assessment following repeat doses as a measure of safety and tolerability | Up to 56 days
  12-lead ECGs will be obtained during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF intervals) at each timepoint
Laboratory parameters assessment following single doses as a measure of safety and tolerability | Up to 61 days
  Laboratory parameters include: hematology, clinical chemistry, and urinalysis
Laboratory parameters following repeat doses as measure of safety and tolerability | Up to 56 days
  Laboratory parameters include: hematology, clinical chemistry, and urinalysis
Number of participants with adverse events following single doses as a measure of safety and tolerability | 33 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact
Number of participants with adverse events following repeat doses as a measure of safety and tolerability | 28 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact

SECONDARY OUTCOMES:
Composite of PK parameters following single doses | PK samples will be collected at pre-dose and 0.2, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose in each of the four dosing session
  PK parameters include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinite]), area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC[0-t]), maximum observed concentration (Cmax), time of occurrence of Cmax (tmax), terminal phase half-life (t1/2)
Composite of PK parameters following repeat doses | Up to 17 days
  PK parameters include: AUC (0-infinite), area under the concentration-time curve over the dosing interval (AUC [0-tau]), AUC (0-t), Cmax, tmax, t1/2 and accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 200181 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200181?search=study&study_ids=200181#rs